CLINICAL TRIAL: NCT04597606
Title: Non-Invasive Ventilation (NIV) Effect on Neurorespiratory Coupling in Chronic Obstructive Pulmonary Disease During Exercise (COPD).
Brief Title: Respiratory Drive Response in COPD Patients During Exercise With Non Invasive Ventilation (NIV).
Acronym: HFNIV
Status: Completed | Type: Observational
Sponsor: Javier Sayas Catalan (Other)
Responsible Party: Sponsor-Investigator, Javier Sayas Catalan, Principal Investigator: Javier Sayas Catalan, Medical Doctor, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Other Study IDs: NIV and HFNC EXERCISE COPD
Record Dates: First submitted 2020-09-18; First posted 2020-10-22 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Noninvasive Ventilation; Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Exercise; Exercise Therapy; Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: All patients will be performed a basal test that consist on continuous cyclergometer exercise, under constant load, with spontaneous breathing, after that the same exercise protocol performed will be carried out under non-invasive ventilation (NIV test). Parameters will be titrated previosuly.
  Finally the patient will perform the same exercise at a constant load under high flow oxygen therapy ( HFNC test).
  Interventions: Other: Exercise with spontaneous ventilation.; Device: Exercise with NIV; Device: Exercise with HFNC

INTERVENTIONS:
Other: Exercise with spontaneous ventilation. — Patients will perform 10 minutes, constant load, exercise in a cycloergometer. To set the load, a baseline incremental effort test will be performed previously (VISIT 1).
  Then, in a separate day (VISIT 2), the subject will perform 10 minutes cycling at the 75% load of that determined as maximum in VISIT 1, at a constant rate of 30 to 35 pedal revolutions per minute, in spontaneous breathing, with low flow oxygen through conventional nasal cannula adjusted to achieve SpO2 between 92to 94%
Device: Exercise with NIV — VISIT 2 Non invasive mask ventilation: parameters will be titrated during a free cycling period at the end of the spontaneous breathing exercise. Then, in a separate day (VISIT 3), with the same constant load, cycling cadence and under NIV, the patient will perform 10 min of cycling.
Device: Exercise with HFNC — With constant flows of 50 lpm and with FiO2 adjusted according to SPO2, to obtain a constant saturation between 92 and 94%. The same pedaling load and frequency will be maintained, with similar variables collected.

SUMMARY:
A constant load exercise during 10 minutes will be performed in a group of Chronic Obstructive Pulmonary Disease patients, in a basal condition (spontaneous breathing); under noninvasive mask ventilation and with high flow nasal cannula. With the aim of reducing dyspnea, increasing exercise tolerance, and unload respiratory muscles, three exercises will be compared in terms of use of respiratory muscles and neural drive measured with paraesternal electromyography.

DETAILED DESCRIPTION:
Exercise in chronic obstructive pulmonary disease is limited by dynamic hyperinflation and respiratory muscle overloadleading to severe dyspnea. During exercise, the increase in neural respiratory drive is notable to match ventilatory demand, correlated with breathlessness. Non-Invasive Ventilation may improve neural respiratory drive uncoupling and exercise tolerance. The aim of this study will be prove if Non-Invasive Ventilation and High flow nasal cannula during exercise reduces neural respiratory drive and improves dyspnea, measured with paraesternal electromyography

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe COPD or cystic fibrosis (with an obstructive pattern and air trapping) on the waiting list for a lung transplant, assessed by the Lung Transplant Unit of the 12 de Octubre University Hospital.
* Diagnostic criteria for COPD according to the GOLD and residual volume greater than 120% of theoretical
* Evidence of developing dynamic air trapping by analyzing flow / volume curves during physical exercise.
* Patients already adapted to home noninvasive mechanical ventilation (NIV) waiting for transplantation.

Exclusion Criteria:

* Presence of comorbidities that limit the patient's physical effort capacity (uncontrolled ischemic heart disease, severe pulmonary hypertension, neuromuscular disease).
* Refusal of treatment with NIV, or inclusion in the study.
* Inability to perform the proposed exercise in basal conditions and with ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recluted from the pneumology outpatient clinic of the Hospital 12 de Octubre
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Changes in Neural ventilator (NVU) (%) | 24 hours, 48 hours, 72 hours
  the peak value (on the baseline) of the maximum muscle activity ( Root mean square EMG value in mV), both diaphragmatic (EMGDimax) and parasternal (EMGparamax) in the máximum intentional ventilation and maximum inspiratory peak (MIP) will be taken. This value will be consider 100% and based on this mean EMG will be calculate for a normalized EMGdi (RMS) and paraesternal in each ventilatory situation (spontaneous ventilation or under NIV). At each effort point (in each minute of the exercise protocol), the relationship between the normalized EMG value (parasternal and Diaphragmatic) and the tidal volume (obtained by integral of flow signal by means of a pneumotachograph connected to the VM -in NIV- or oronasal hermetic mask -in Vesp). To facilitate the interpretation of the expired TV, the mask without leakage will be used with the intentional leak connected in the circuit, before the pneumotachograph.

SECONDARY OUTCOMES:
Borg Scale Dyspnea evolution (points) | Basal value at day 1 and every 60 seconds during the exercise
  Degree of dyspnea will be determined by this validated scale with a result between 1 and 10 points.0: Not at all 0.5: Very, very light (hardly noticeable) 1: Very light, 2: Light, 3: Moderate , 4: Somewhat intense, 5: Intense, 6: Between 5 and 7, 7: Very intense, 8: Between 7 and 9, 9: Very, very intense (almost maximum ), 10: Maximum
Borg Scale Dyspnea evolution (points) | 24 hours later than day 1 (day 2) during the exercise every 60 seconds
  Degree of dyspnea will be determined by this validated scale with a result between 1 and 10 points.0: Not at all 0.5: Very, very light (hardly noticeable) 1: Very light, 2: Light, 3: Moderate , 4: Somewhat intense, 5: Intense, 6: Between 5 and 7, 7: Very intense, 8: Between 7 and 9, 9: Very, very intense (almost maximum ), 10: Maximum
Borg Scale Dyspnea evolution (points) | 48 hours later than day 1 (day 3) during the exercise every 60 seconds
  Degree of dyspnea will be determined by this validated scale with a result between 1 and 10 points.0: Not at all 0.5: Very, very light (hardly noticeable) 1: Very light, 2: Light, 3: Moderate , 4: Somewhat intense, 5: Intense, 6: Between 5 and 7, 7: Very intense, 8: Between 7 and 9, 9: Very, very intense (almost maximum ), 10: Maximum
Borg Scale Dyspnea evolution (points) | 72 hours later than day 1 (day 4) during the exercise every 60 seconds
  Degree of dyspnea will be determined by this validated scale with a result between 1 and 10 points.0: Not at all 0.5: Very, very light (hardly noticeable) 1: Very light, 2: Light, 3: Moderate , 4: Somewhat intense, 5: Intense, 6: Between 5 and 7, 7: Very intense, 8: Between 7 and 9, 9: Very, very intense (almost maximum ), 10: Maximum
Transcutaneous pCO2 Final - inicial (mmHg) | Basal value at day 1 during the exercise
  Transcutaneous monitor uses a noninvasive technique to measure the skin-surface partial pressure of carbon dioxide (PtcCO2)
Transcutaneous pCO2 Final - inicial (mmHg) | During the exercise at day 2 ( 24 hours later than day 1)
  Transcutaneous monitor uses a noninvasive technique to measure the skin-surface partial pressure of carbon dioxide (PtcCO2)
Transcutaneous pCO2 Final - inicial (mmHg) | During the exercise at day 3 (48 hours later than day 1)
  Transcutaneous monitor uses a noninvasive technique to measure the skin-surface partial pressure of carbon dioxide (PtcCO2)
Transcutaneous pCO2 Final - inicial (mmHg) | During the exercise at day 4 (72 hours later than day 1 )
  Transcutaneous monitor uses a noninvasive technique to measure the skin-surface partial pressure of carbon dioxide (PtcCO2)
Total Training time (pedaling, minutes) | During the exercise at day 2 ( 24 hours later than day 1)
  Total Time that the patient remains pedaling
Total Training time (pedaling, minutes) | During the exercise at day 3 ( 48 hours later than day 1)
  Total Time that the patient remains pedaling
Total Training time (pedaling, minutes) | During the exercise at day 4 ( 72 hours later than day 1)
  Total Time that the patient remains pedaling
Stops (n) | During the exercise at day 2 ( 24 hours later than day 1)
  Number of stops that the patient performs during the test
Stops (n) | During the exercise at day 3 ( 48 hours later than day 1)
  Number of stops that the patient performs during the test
Stops (n) | During the exercise at day 4 ( 72 hours later than day 1)
  Number of stops that the patient performs during the test
Ineffective efforts % | During the exercise at day 2 ( 24 hours later than day 1)
  Porcentage of ineffective efforts during the exercise
Ineffective efforts % | During the exercise at day 3 ( 48 hours later than day 1)
  Porcentage of ineffective efforts during the exercise
Ineffective efforts % | During the exercise at day 4 ( 72 hours later than day 1)
  Porcentage of ineffective efforts during the exercise

CONTACTS AND LOCATIONS:
Overall Officials: Javier Sayas, Principal Investigator — Hospital 12 de OCtubre
Locations (1):
- Javier Sayas Catalan, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sayas J, Lalmolda C, Corral M, Florez P, Hernandez-Voth A, Janssens JP, Rabec C, Langevin B, Lofaso F, Carlucci A, Llontop C, Winck JC, Bermejo JG, Lujan M. Measurement of thoraco-abdominal synchrony using respiratory inductance plethysmography: technical aspects and a proposal to overcome its limitations. Expert Rev Respir Med. 2024 Mar-Apr;18(3-4):227-236. doi: 10.1080/17476348.2024.2363058. Epub 2024 Jun 7. PMID 38829281

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT04597606/Prot_SAP_ICF_000.pdf